CLINICAL TRIAL: NCT01509924
Title: Cognitive and Physical Functions in Patients With TIA. A Randomized Controlled Trial of Physical Activity on Prescription up to One Year After the Event
Brief Title: Cognitive and Physical Functions in Patients With Transient Ischemic Attack. A Randomized Controlled Trial of Physical Activity on Prescription up to One Year After the Event
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tiohundra AB (Industry)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Carina Moren, Principal Investigator, Tiohundra AB
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tiohundra
Record Dates: First submitted 2011-06-07; First posted 2012-01-13 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Ischemic Attack, Transient
Keywords: Walking capacity; Mental Fatigue; Quality of Life; Cognition; Motor activity; Exercise
MeSH Terms: conditions — Ischemic Attack, Transient; Mental Fatigue; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Physical activity on Prescription (PaP) (Experimental): Intervention group receives a PaP for 12 month.
  Interventions: Other: Physical activation on Prescription
- Control Group (No Intervention): The control group has the same monitoring as the experimental group but receives no PaP.
- Cognitiv function in patients with TIA (No Intervention): Before discharged from hospital cognitive function is assessed. At the first visit the patients fill in a self assessment questionnaire for mental fatigue.
  If impaired at the previous assessment cognitive function will be assessed at 3, 6 and 12 month.
- Controlgroup Cognitive function (No Intervention): In order to determine whether hospitalization in itself is associated with transient impaired cognition, a comparison group will be included. The comparison group will consist of patients with angina pectoris consecutively admitted to the Norrtälje Hospital. The patients with angina pectoris will be age and sex matched with the patients with TIA and assessed for cognitive function when their angina symptoms have subsided.

INTERVENTIONS:
Other: Physical activation on Prescription — The advice on physical activity is patient oriented and based on FYSS (FYSS is a information bank that summarizes the up-to-date scientific knowledge on how to prevent and treat various diseases and conditions using physical activity). An individual prescription on physical activity is issued. The prescription form reminds of an ordinary drug prescription and provides specified types of physical activities including intensity, frequency and duration of the respective activities. The prescribed physical activity could be either self-monitored or organized by public physical activity organizations.
  Other Names: PaP
  Arms: Physical activity on Prescription (PaP)

SUMMARY:
The purpose of this study is to determine whether Physical Activation on Prescription can help patients with TIA to become more physically active.

One group will receives Physical Activation on Prescription (PaP)and the other group will receives usual care.

And to identify if persons with TIA presents with cognitive impairments.

DETAILED DESCRIPTION:
Transient ischemic attack (TIA) is a transient episode of neurologic dysfunction caused by ischemia, i.e. loss of blood flow. The symptoms of a TIA typically resolve within 24 hours. Attacks lasting more than 30 minutes are unusual. TIAs and strokes present with the same symptoms such as sudden weakness, numbness, sudden dimming or loss of vision, aphasia, slurred speech, facial palsy and mental impairments. Subtle problems with cognitive functions and fatigue may not always be addressed before discharge. However, even subtle mental impairments are important to identify, given the problems they might pose.

ELIGIBILITY:
Inclusion Criteria:

* Understand Swedish language (also in and writing), living in Norrtälje community,
* To participate in the assessment of cognitive function: no known cognitive impairments before the TIA event and history of stroke.

Exclusion Criteria:

* Presence of contraindications to exercise, and no history of stroke

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-05; Primary Completion 2015-04 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Change in Physical activity over time | at discharge from hospital, 3, 6 and 12 month after the event
  Physical activity measured with accelerometer (Time frame: Baseline, 3, 6, and 12 month).

SECONDARY OUTCOMES:
Change in Cognition and Mental Fatigue | All measures at baseline 3, 6 and 12 month after the event
  Change in mental conditions over time measured with self report of mental fatigue and related symptoms. This is a scale with 7 different steps for graduate mental fatigue. Less points indicate less mental fatigue.
Change in 6 MWT | 3, 6 and 12 months
  Change in Walking endurance measured in 3, 6, 12 month measured with 6 MWT (six minutes Walking Test).
Change in self reported stages of change | 3, 6, 12 months
  A self reported questionnaire that measures willingness to changes in physical activity over time. The scale has different levels of willingness for changes in physical activity.
Change from baseline in systolic blood pressure at 12 months | 3, 6, 12 months
BMI | 12 months
  Body Mass Index is measured at the start and at the end of the study
Change in mental capacity over a period of time | 3, 6,12 months
  Change in mental capacity measured with a assessment called Cognistat that indicates four different levels of mental capacity.
Change in mental capacity over a period of time | 3, 6, 12 months
  Change in mental capacity measured with a assessment called Cognistat that indicates four different levels of mental capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Disa Sommerfeld, Study Director — Karolinska Institutet
Locations (1):
- Tiohundra, Norrtälje, Stockholms Läns Landsting, Sweden